CLINICAL TRIAL: NCT05390411
Title: Seeking Objectivity in Allocation of Advanced Heart Failure (SOCIAL HF) Therapies Trial
Acronym: SOCIAL HF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Khadijah Breathett, MD, MS, FACC, FAHA, FHFSA, tenured Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13943; R56HL159216 (NIH); R01HL159216 (NIH)
Record Dates: First submitted 2022-03-21; First posted 2022-05-25 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-06

CONDITIONS: Implementation Science; Heart Transplant; Decision Making
Keywords: Healthcare Disparities

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controlled cluster trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Sites (No Intervention): No Intervention
- Sites Randomized to SOCIAL HF (Experimental): SOCIAL HF is composed of evidence-based disparities reduction training, employment of objective measures of social support, and changes to facilitate group dynamics.
  Interventions: Behavioral: SOCIAL HF

INTERVENTIONS:
Behavioral: SOCIAL HF — participate in SOCIAL HF training
  Arms: Sites Randomized to SOCIAL HF

SUMMARY:
The primary goal of this study is to assess real-world effectiveness and implementation of an evidence-based multi-component strategy to reduce disparities in the allocation rate of advanced heart failure therapies, heart transplants and ventricular assist devices. This study proposes to implement evidence-based strategies that reduce unequal and unethical decision-making towards patients, replace subjective evaluations with objective criteria, and improve group dynamics in a randomized cluster trial. Our rigorously designed trial will inform national guidelines for advanced heart failure therapy allocation, and data are likely to be generalizable to other organ replacement treatments and advanced chronic disease decision-making processes across populations.

DETAILED DESCRIPTION:
Standardized protocols can reduce the impact of unfair and unequal treatment but are underused. Since the Institute of Medicine's report, "Unequal Treatment", multiple studies have confirmed that standardization of decision-making processes reduces unequal treatment, but unequal and unethical perceptions in decision-making in the allocation of advanced therapies has not been addressed. Using an evidence-based framework for behavior change [Capability, Opportunity, and Motivation for Behavior Change/Behavior Change Wheel (COM-B/BCW)], we developed a standardized protocol strategy, Seeking Objectivity in Allocation of Advanced Heart Failure (SOCIAL HF), that addresses the most significant barriers to equality in advanced therapies: 1) unequal and unethical perceptions that influence decision-making, 2) subjectivity in evaluation of social support and adherence, and 3) poor group dynamics. Thus, SOCIAL HF includes: 1) evidence-based training to reduce disparities tailored for HF, 2) restriction to objective evaluations of social support and adherence, and 3) environmental restructuring and modeling of meeting settings to include anonymous electronic voting and more fair-minded seating arrangement. In complex decision-making that includes individuals and groups, our standardized protocol strategy, SOCIAL HF, has the greatest likelihood of reducing health disparities in advanced HF. Our goal is to assess real-world effectiveness (Aim 1) and implementation (Aim 2) of SOCIAL HF for allocation of advanced HF therapies, heart transplant and ventricular assist device implantation. As a type 2 effectiveness-implementation hybrid study, we will use a cluster randomized design to test the effectiveness of SOCIAL HF strategy. We will evaluate implementation of SOCIAL HF across study sites using mixed-methods to learn optimal implementation strategies to reduce disparities in accessing life-saving therapies. We will use normalization process theory to evaluate how SOCIAL HF affects processes and outcomes important to advanced HF centers (e.g. fidelity/variation). We will use RE-AIM framework (reach, effectiveness, adoption, implementation, and maintenance) to evaluate factors that promote reach and adoption and resources needed for implementation. We have the relationships, infrastructure, and expertise to execute this project; our multidisciplinary team includes experts in HF, evidence-based training in reducing unequal and unethical perceptions in decision-making, clinical trials, mixed-methods, and implementation science.

ELIGIBILITY:
Inclusion Criteria:

1. Active United Network for Organ Sharing heart transplant and ventricular assist device center
2. Centers that routinely evaluate at least 50 minoritized racial/ethnic patients and 50 women for advanced heart failure therapies (heart transplant and ventricular assist device) over 2 years
3. Advanced therapy professionals from participating centers (i.e., coordinators, physicians, pharmacists, nurses, social workers)
4. Participants for the interview portion will be a subset of otherwise eligible advanced therapy professionals who are included on selection meeting attendance sheets at an included center

Exclusion Criteria:

1. Centers unable to fully participate in the training and evaluation measures
2. If the center ceases to be an active heart failure/transplant center

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1463 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of evaluated minoritized racial/ethnic patients and women patients receiving advanced therapies. | Up to 2 years
Change in SOCIAL HF fidelity from time of training completion (month 2) to time study target has been reached (up to 2 years) and 6 months after reaching study target (up to 2.5 years) | Month 2, up to 2 years, and up to 2.5 years
  Evaluated as barriers, facilitators, and variability in adoption, reach, implementation and maintenance through structured interviews.
  Study target is defined as time 50 patients of color and 50 women have been evaluated for advanced heart failure therapies per center.

SECONDARY OUTCOMES:
Change from baseline knowledge, attitudes, and self-reported behavior change among clinicians at 2 months and time at which study target has been reached (up to 2 years) | Baseline, 2 months, and up to 2 years
  Multiple survey responses by participants will indicate knowledge, attitudes, and self-reported behavior changes over time.
  Study target is defined as time 50 patients of color and 50 women have been evaluated for advanced heart failure therapies.
Discussion themes during allocation meetings across patient race/ethnicity and sex | Baseline, 2 months, and up to 2 years
  Transcriptions of meetings will be qualitatively evaluated over time.
Change from baseline sum group function scores at 2 months and time at which study target has been reached (up to 2 years) | Baseline, 2 months, and up to 2 years
  The de Groot Critically Reflective Diagnoses protocol objectively measures categories associated with group function including challenging groupthink, critical opinion sharing, research utilization, openness to mistakes, asking and giving feedback, and experimentation. Each category is scaled from 1-4 (high-low), 1 = demonstrating interaction and reflection, 2 = reflective on an individual basis, 3 = non-reflective and non-interactive, and 4 = restricted.
  Study target is defined as time 50 patients of color and 50 women have been evaluated for advanced heart failure therapies per center.
Adoption of SOCIAL HF | 2 months
  Proportion of eligible advanced therapy professionals who participate in training
Reach of SOCIAL HF | From 2 months up to 2 years
  Proportion of patients evaluated using any parts of SOCIAL HF
Implementation of SOCIAL HF | From 2 months up to 2 years
  Proportion of patients evaluated using all parts of SOCIAL HF

CONTACTS AND LOCATIONS:
Overall Officials: Khadijah Breathett, MD, MS, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Reporter — https://reporter.nih.gov/search/PL_QHU4f3EadVajKcfIy9A/project-details/10474768
- See also: NIH Reporter — https://reporter.nih.gov/search/PL_QHU4f3EadVajKcfIy9A/project-details/10440891